CLINICAL TRIAL: NCT01431261
Title: Neck Exercises, Physical and Cognitive Behavioural Graded Activity as a Treatment for Adult Whiplash Patients With Chronic Neck Pain
Brief Title: Neck Exercises, Training and Pain Management as a Treatment for Whiplash Patients With Chronic Neck Pain
Acronym: WADNECXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); Association of Danish Physiotherapists (Other)
Responsible Party: Principal Investigator, Inge Ris Hansen, PhD. student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WADNECXT
Record Dates: First submitted 2011-08-30; First posted 2011-09-09 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Neck Pain; Chronic Pain Syndrome
Keywords: Chronic neck pain; Whiplash; Whiplash Associated Disorders; Chronic Pain; Neck exercises; Training; Pacing; Patient Education; Pain Management; Whiplash Injuries; Musculoskeletal
MeSH Terms: conditions — Neck Pain; Whiplash Injuries; Chronic Pain; Agnosia | interventions — Educational Status; Pain Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain Management + Training (Active Comparator): Education in pain management strategies and treatment sessions including instructions in neck exercises and aerobic training
  Interventions: Other: Education and training
- Pain Management (Active Comparator): Education in pain management strategies
  Interventions: Behavioral: Pain management

INTERVENTIONS:
Other: Education and training — Educational sessions in pain management 4 times and treatment sessions including instructions in training and specific exercises 8 times
  Arms: Pain Management + Training
Behavioral: Pain management — Educational sessions in pain management 4 times
  Arms: Pain Management

SUMMARY:
The purpose of this study is to test whether a physiotherapy intervention containing pain management, general training and specific neck exercises can improve function for patients with chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is widespread problem. The prevalence of neck pain in the Scandinavian countries is 36%. Of the working population the prevalence of chronic neck pain is 10 - 20%.The National Board of Health estimates that 5-6000 subjects per year in Denmark are involved in a traffic accident evoking whiplash-induced chronic neck pain. The main problems for patients with chronic neck pain are cervical dysfunction, reduced neck mobility and stability in addition to local and possibly generalised pain Besides chronic neck pain, patients may suffer from poor pain coping strategies and physical inactivity which influences physical function, general health and causes a poor quality of life.

Physical training including specific exercises targeting the deep postural muscles of the spine is effective in reducing neck pain for patients with chronic neck pain. Physical behavioural graded activity is a treatment approach with focus on increasing general physical fitness, reducing fear of movements and increasing psychological function. Educational sessions, where the focus is on understanding complex chronic pain mechanisms and development of appropriate pain coping and/or cognitive behavioural strategies have shown reduced general pain.

Thus this project is formulated on the expectation that rehabilitation of patients with chronic neck pain after a whiplash accident must target cervical dysfunctions, training of physical function and the understanding and management of chronic pain in a combined therapy approach.

The study is designed as a randomized control study including 200 patients. All participate in the educational sessions. The training group receives on top of that instruction in specific neck exercises and general training.

ELIGIBILITY:
Inclusion Criteria:

* chronic neck pain for at least 6 months
* reduced physical neck function (NDI minimum 10)
* pain primarily in the neck region,
* finished any medical /radiological examinations
* able to read and understand Danish and
* able to participate in the exercise program.

Exclusion Criteria:

* radiculopathies upper extremity
* neurological deficits
* in a process of examining for unknown pathology,
* experimental medical treatment,
* being in a unstable social situation
* pregnancy
* fractures
* suffering from depression
* other known coexisting medical conditions which would severely restrict participation in the exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study Short Form 36 (SF36) - Physical Component Summary (PCS) | 12 months

SECONDARY OUTCOMES:
craniocervical flexion test | 12 months
  test for the deep cervical flexor muscles
cervical range of motion | 12 months
neck positioning test | 12 months
  neck joint position error test and gaze stability test
Self-rated measure Global Perceived Effect | 12 months
  questionnaire
Neck Disability Index | 12 months
  questionnaire
Pain Bothersomeness | 12 months
  questionnaire
Pain Specific Functioning Scale | 4 months and 12 months
  questionnaire
TAMPA scale of Kinesiophobia | 12 months
  questionnaire
Impact of Event scale | 12 months
  questionnaire
Euroqol-5D | 12 months
  questionnaire
Mechanical allodynia | 12 months
  Pressure pain treshold for selected points

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Juul-Kristensen, ph.d., Study Chair — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Research Unit for Musculoskeletal Function and Physiotherapy, Institute of Sports Science and Clinical Biomechanics, Odense, Denmark

REFERENCES:
- [Derived] Ris I, Juul-Kristensen B, Boyle E, Kongsted A, Manniche C, Sogaard K. Chronic neck pain patients with traumatic or non-traumatic onset: Differences in characteristics. A cross-sectional study. Scand J Pain. 2017 Jan;14:1-8. doi: 10.1016/j.sjpain.2016.08.008. Epub 2016 Oct 12. PMID 28850421
- [Derived] Ris I, Sogaard K, Gram B, Agerbo K, Boyle E, Juul-Kristensen B. Does a combination of physical training, specific exercises and pain education improve health-related quality of life in patients with chronic neck pain? A randomised control trial with a 4-month follow up. Man Ther. 2016 Dec;26:132-140. doi: 10.1016/j.math.2016.08.004. Epub 2016 Aug 20. PMID 27598552
- [Derived] Hansen IR, Sogaard K, Christensen R, Thomsen B, Manniche C, Juul-Kristensen B. Neck exercises, physical and cognitive behavioural-graded activity as a treatment for adult whiplash patients with chronic neck pain: design of a randomised controlled trial. BMC Musculoskelet Disord. 2011 Dec 2;12:274. doi: 10.1186/1471-2474-12-274. PMID 22136113
- See also: University of Southern Denmark — http://www.sdu.dk